CLINICAL TRIAL: NCT02695186
Title: Markers of Oxidative Stress and Inflammation in Patients With Intestinal Metaplasia and Metabolic Syndrome
Brief Title: Oxidative Stress in Intestinal Metaplasia and Metabolic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Hospital of Filiates (Other Government)
Collaborators: University of Ioannina (Other)
Responsible Party: Sponsor
Other Study IDs: 1/21/01/2016
Record Dates: First submitted 2016-02-19; First posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Intestinal Metaplasia; Metabolic Syndrome; Oxidative Stress; Inflammatory Response
Keywords: Intestinal metaplasia; Metabolic syndrome; Oxidative stress
MeSH Terms: conditions — Metabolic Syndrome | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- A/IM alone: Patients with intestinal metaplasia who undergo gastroscopy and blood sample analysis
  Interventions: Procedure: Gastroscopy
- B/IM and MS: Patients with intestinal metaplasia and metabolic syndrome who undergo gastroscopy and blood sample analysis
  Interventions: Procedure: Gastroscopy
- C/Healthy controls: Healthy controls without intestinal metaplasia or metabolic syndrome who undergo gastroscopy and blood sample analysis
  Interventions: Procedure: Gastroscopy

INTERVENTIONS:
Procedure: Gastroscopy — Gastroscopy and biopsies, as well as blood sample collection

SUMMARY:
Intestinal metaplasia is generally considered a precancerous lesion. Although it is associated with a very small increase of gastric cancer risk, European Endoscopic Society and other European academic companies highlighted the increased risk of cancer in patients with gastric atrophy and IM and the need for staging in cases with high-grade dysplasia.

The production of ROS in the gastrointestinal tract (GI) and their role in the pathophysiology and pathogenesis of gastrointestinal diseases have not been studied sufficiently. In the plasma of patients, in the context of the sequence gastro oesophageal reflux-oesophagitis-metaplasia-dysplasia-adenocarcinoma, have been found simultaneous formation of DNA adducts and increased myeloperoxidase concentration, which are associated with oxidative stress, decreased antioxidant capacity (decreased glutathione concentration).These findings support the role of oxidative stress in the pathogenesis and malignant transformation.

Metabolic Syndrome (MS) has been recognized as a pro-inflammatory, pro-coagulant state associated with increased levels of C reactive protein (CRP), interleukin (IL) 6 and plasminogen activator inhibitor (PAI) 1. It has been reported that the inflammatory and the pro thrombotic markers, which are associated with increased risk for cardiovascular disease and DM2, represent only a part of the relationship between IM and cardiovascular mortality.

Several factors influence the pathogenesis of MS, as the pro-oxidant condition of such patients may increase the risk for developing symptoms and related chronic diseases such as DM2. Although the exact contribution of oxidative stress on every pathologic condition included in MS is difficult to determine definitively, it is certain that oxidative stress is particularly high in the MS.

Regarding the relationship between MS and GI diseases, studies have reported that patients with MS are almost twice at risk for developing Barrett's esophagus.The relationship between MS, gastro-esophageal reflux disease (GERD), and the development of IM also requires well designed prospective studies. It seems however, to be a correlation between obesity and GERD, as well as between obesity and gastric adenocarcinoma

DETAILED DESCRIPTION:
INTRODUCTION:

Intestinal metaplasia (IM) is considered a precancerous lesion and is associated with a very small increase of gastric cancer risk. Generally there are no widely accepted guidelines on the IM management. Recently, the European Endoscopic Society and other European academic companies have developed evidence-based guidelines for the management of patients with IM. These instructions highlighted the increased risk of cancer in patients with gastric atrophy and IM and the need for staging in cases with high-grade dysplasia. Risk factors for IM include infection with Helicobacter pylori, high NaCl intake, smoking, alcohol consumption and chronic bile reflux. The four steps sequence of the events for the development of the intestinal type gastric adenocarcinoma include: Non-atrophic gastritis, multifocal atrophic gastritis, IM, and dysplasia.

Reactive oxygen species (ROS) are produced as by-products of the normal metabolism of the cell. ROS are generated in response to ultraviolet radiation, smoking, alcohol, nonsteroidal anti-inflammatories, ischemia-reperfusion, chronic infections and chronic inflammatory disorders. Disruption of the normal homeostasis of the cell, due to changes in redox homeostasis can lead to the development of cardiovascular diseases, neurodegenerative diseases and cancer. The production of ROS in the gastrointestinal tract (GI) and their role in the pathophysiology and pathogenesis of gastrointestinal diseases have not been studied sufficiently. Despite the protective barrier provided by the digestive mucosa, different molecules which may be present in the content of GI,as well as various pathogens can cause oxidative damage and inflammatory response in the intestinal mucosa and the immune cells. Pathogenesis of various GI diseases, including ulcerative lesions, cancer, and inflammatory bowel diseases are attributable in part to oxidative stress. In the plasma of patients, in the context of the sequence gastro oesophageal reflux-oesophagitis-metaplasia-dysplasia-adenocarcinoma, have been found simultaneous formation of DNA adducts and increased myeloperoxidase concentration, which are associated with oxidative stress, decreased antioxidant capacity (decreased glutathione concentration).These findings support the role of oxidative stress in the pathogenesis and malignant transformation.

On the other hand, since chronic inflammation has been recognized as an important risk factor for the development of GI tumors, the underlying molecular mechanisms have been studied extensively. Chronic inflammation may induce cell mutations and promote malignant transformation in normal cells of the GI mucosa. The inflammatory reaction generated during carcinogenesis involves the formation of reactive oxygen and nitrogen species (ROS and RNS) derived from mononuclear phagocytes and lymphocytes, as well as the development of immune response, and the production of pro-inflammatory cytokines. Nuclear factor-κB (NF-κB) is considered as the main mediator of the immune response. The activation of NF-κB through phosphorylation leads to translocation of NF-κB in the nucleus, where regulates the transcription of several pro-inflammatory cytokines and chemokines. Furthermore, chronic inflammation can create the appropriate conditions for genomic and epigenetic changes.

Obesity, particularly abdominal obesity, is associated with insulin resistance in the peripheral tissues and abnormal fatty acid metabolism, often leading to type 2 diabetes mellitus (DM2) development. Insulin resistance, hyperinsulinemia, hypoglycemia and cytokine production by adipocytes (adipokines) can also result in endothelial dysfunction, disorders of the lipid profile, hypertension and vascular inflammation, which promote the development of atherosclerotic cardiovascular disease. In patients with coexistence of metabolic risk factors for DM2 and cardiovascular disease (abdominal obesity, hyperglycemia, dyslipidemia and hypertension) suggested the existence of "metabolic syndrome". Metabolic Syndrome (MS) has been recognized as a pro-inflammatory, pro-coagulant state associated with increased levels of C reactive protein (CRP), interleukin (IL) 6 and plasminogen activator inhibitor (PAI) 1. It has been reported that the inflammatory and the pro thrombotic markers, which are associated with increased risk for cardiovascular disease and DM2, represent only a part of the relationship between IM and cardiovascular mortality. Furthermore, no causal relationship between increased levels of CRP levels and MS incidence has been found. The value of several markers for the monitoring of patients with MS remain uncertain.The use of these markers should be made for clinical purposes only, with respect to the determination of cardiovascular risk assessment. The guidelines of the Centers for Disease Control and Prevention (CDC) emphasize that the analysis of CRP still belongs to the optional tests, because the power as an independent predictive remains uncertain.

Several factors influence the pathogenesis of MS, as the pro-oxidant condition of such patients may increase the risk for developing symptoms and related chronic diseases such as DM2. The reduction of antioxidant capacity in individuals with IM can be explained by the concomitant overproduction of ROS and their metabolites (d-ROMS), the decreased activity of the enzymes that neutralize ROS (SOD, CAT and GPx) and reduction of other antioxidant systems, such as PON1 activity. Recently, γGT has been suggested as a promising biomarker for the diagnosis of MS, and its levels in serum may reflect the response to oxidative stress.

Moreover, the correlation between the SOD and the various active moieties in MS may indicate that the SOD activity could be a better biomarker of oxidative stress in these patients. The measurement of the SOD activity could be used as a predictive tool for determining the extent of the underlying oxidative stress in the disease. These findings suggest that the study of the oxidative state in the earlier phases of MS may be the starting point for understanding the pathways that contribute to the progress of the MS and its subsequent complications. Although the exact contribution of oxidative stress on every pathologic condition included in MS is difficult to determine definitively, it is certain that oxidative stress is particularly high in the MS. It seems that increased oxidative stress is the main mechanism behind the increased tendency to develop cardiovascular disease, greater severity of cardiovascular disease in younger people and poorer treatment outcomes.

Regarding the relationship between MS and GI diseases, studies have reported that patients with MS are almost twice at risk for developing Barrett's esophagus. If these findings will be confirmed in prospective studies, patients with MS could form a high-risk group for developing Barett's esophagus and esophageal adenocarcinoma. The prevalence of MS concerning the development of Barett's esophagus and particularly the relationship between the length of damage and changes in the levels of leptin, insulin and proinflammatory markers, indicate that the changes caused by the development of Barrett's esophagus are constant and are affected by metabolic changes caused by adipokines and cytokines. The relationship between MS, gastro-esophageal reflux disease (GERD), and the development of IM also requires well designed prospective studies. It seems however, to be a correlation between obesity and GERD, as well as between obesity and gastric adenocarcinoma.

AIM OF THE STUDY:

This study aim the analysis of oxidative stress markers and markers of inflammation in patients with IM and MS, patients with IM alone, and healthy volunteers, as well as the impact of therapeutic protocols, and the association of the markers with the extension of the lesion.

MATERIALS AND METHODS:

A group of patients with IM and MS, a group of patients with IM alone, and a group of healthy volunteers. Every group of patients will be divided in subgroups based on age and gender.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of metabolic syndrome, Must be able to undergo gastroscopy,
* Must be >25 and <75 years old

Exclusion Criteria:

* Autoimmune diseases, Malignancy, Chronic kidney disease, Type 2 diabetes complications

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A group of patients with IM and MS, a group of patients with IM alone, and a group of healthy volunteers. Every group of patients will be divided in subgroups based on age and gender.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
8-epiPGF2α (pg/ml) | Baseline
  Marker of lipid peroxidation
8-OHG (ng/ml) | Baseline
  Marker of RNA oxidation
Total antioxidant capacity (TAC) (mM) | Baseline
  Measurement of antioxidant concentration (Uric acid, ascorbic acid, Vitamin E, BHT, Triolox, GSH, BSA/PBS)
Total cholesterol (mg/dl) | Baseline
LDL-C (mg/dL) | Baseline
HDL-C (mg/dL) | Baseline
Triglycerides (TRG) (mg/dL) | Baseline
BMI (kg/height2) | Baseline
Plasma glucose (mg/dL) | Baseline
Plasma glycated hemoglobin A1c (%) | Baseline

SECONDARY OUTCOMES:
Correlation between markers of oxidative stress and extension of the gastric lesion | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Pappas-Gogos, MD, MSc, Principal Investigator — Filiates General Hospital
Locations (1):
- General Hospital of Filiates, Filiátes, Epirus, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Correa P, Piazuelo MB, Wilson KT. Pathology of gastric intestinal metaplasia: clinical implications. Am J Gastroenterol. 2010 Mar;105(3):493-8. doi: 10.1038/ajg.2009.728. No abstract available. PMID 20203636
- [Background] Chandrasoma P, Wickramasinghe K, Ma Y, DeMeester T. Is intestinal metaplasia a necessary precursor lesion for adenocarcinomas of the distal esophagus, gastroesophageal junction and gastric cardia? Dis Esophagus. 2007;20(1):36-41. doi: 10.1111/j.1442-2050.2007.00638.x. PMID 17227308
- [Background] Bhattacharyya A, Chattopadhyay R, Mitra S, Crowe SE. Oxidative stress: an essential factor in the pathogenesis of gastrointestinal mucosal diseases. Physiol Rev. 2014 Apr;94(2):329-54. doi: 10.1152/physrev.00040.2012. PMID 24692350
- [Background] Sihvo EI, Salminen JT, Rantanen TK, Ramo OJ, Ahotupa M, Farkkila M, Auvinen MI, Salo JA. Oxidative stress has a role in malignant transformation in Barrett's oesophagus. Int J Cancer. 2002 Dec 20;102(6):551-5. doi: 10.1002/ijc.10755. PMID 12447994
- [Background] Meigs JB. Invited commentary: insulin resistance syndrome? Syndrome X? Multiple metabolic syndrome? A syndrome at all? Factor analysis reveals patterns in the fabric of correlated metabolic risk factors. Am J Epidemiol. 2000 Nov 15;152(10):908-11; discussion 912. doi: 10.1093/aje/152.10.908. PMID 11092432
- [Background] Hutcheson R, Rocic P. The metabolic syndrome, oxidative stress, environment, and cardiovascular disease: the great exploration. Exp Diabetes Res. 2012;2012:271028. doi: 10.1155/2012/271028. Epub 2012 Jul 9. PMID 22829804